CLINICAL TRIAL: NCT05169710
Title: A Multi-region, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study Evaluating SEP-4199 Controlled Release (CR) for the Treatment of Major Depressive Episode Associated With Bipolar I Disorder (Bipolar I Depression)
Brief Title: A Clinical Study of an Investigational Drug for the Treatment of Major Depressive Episode Associated With Bipolar I Disorder.
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Company decided not to move forward with further accrual.
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SEP380-301; 2021-002126-24 (EudraCT Number); jRCT2031210559 (Registry Identifier: Japan Registry for Clincal Trials)
Record Dates: First submitted 2021-12-13; First posted 2021-12-27 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-09

CONDITIONS: Depressive Episodes, Bipolar I Depression
Keywords: Depression, Depressive episode, Bipolar, Bipolar 1, Bipolar 1 depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled, Parallel-Group
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SEP-4199 CR 200 mg (Experimental): SEP-4199 CR 200 mg/day
  Interventions: Drug: SEP-4199 CR 200 mg
- SEP-4199 CR 400 mg (Experimental): SEP-4199 CR 400 mg/day
  Interventions: Drug: SEP-4199 CR 400 mg
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SEP-4199 CR 200 mg — SEP-4199 CR 200 mg Tablet (supplied in one 200mg tablet and one placebo tablet)
  Arms: SEP-4199 CR 200 mg
Drug: SEP-4199 CR 400 mg — SEP-4199 CR 400 mg tablet (supplied in two 200mg tablets)
  Arms: SEP-4199 CR 400 mg
Drug: Placebo — Placebo tablet (supplied in two tablets)
  Arms: Placebo

SUMMARY:
A clinical trial to study the efficacy and safety of an investigational drug in people with major depressive episodes associated with with Bipolar I disorder (bipolar I depression) Participants in the study will either receive the drug being studied or a placebo. The study will be conducted in approximately 90 sites in North America, Europe, Latin America and Japan. It will be have both male and female participants ages 18-65. Participation in the study will be approximately 10 weeks.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, placebo-controlled, parallel-group study designed to evaluate the efficacy, safety, and tolerability of treatment with SEP-4199 CR at fixed doses of 200 mg/day or 400 mg/day compared with placebo for the treatment of major depressive episode associated with bipolar I disorder (bipolar I depression). The study is projected to randomize approximately 522 subjects inNorth America, Japan, Europe and Latin America, to SEP-4199 CR 200 mg/day, SEP-4199 CR 400 mg/day, and placebo treatment groups in a 1:1:1 ratio

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria (not all inclusive):

* Subject provides written informed consent and is willing and able to comply with the protocol in the opinion of the Investigator.
* Subject is 18 to 65 years of age, inclusive, at the time of informed consent.
* Subject meets DSM-5 criteria, based on the SCID-5-CT, for bipolar I disorder, current episode depressed with or without rapid cycling disease course (≥ 4 episodes of mood disturbance but < 8 episodes in the previous 12 months) with or without psychotic features.
* Subject's current major depressive episode is ≥ 4 weeks and less than 12 months in duration at Screening.
* Subject has a MADRS total score ≥ 22 at both Screening and Baseline.
* Subject has a CGI-BP-S depression score ≥ 4 at both Screening and Baseline.
* Subject has a YMRS total score ≤ 12 at both Screening and Baseline.
* Subject is in good physical health, based on medical history, physical examination, neurological examination, vital signs, ECGs, and results of clinical laboratory tests (hematology, chemistry, and urinalysis).

Exclusion Criteria:

Exclusion Criteria (not all inclusive):

* Subject currently has any DSM-5 defined psychiatric diagnosis other than bipolar I disorder that was the primary focus of treatment, or is currently being treated with concomitant medication
* Subject has a lifetime history of, or symptoms consistent with, schizophrenia, schizoaffective disorder, or a major psychiatric diagnosis other than bipolar I disorder that is judged to pose risk to the study scientific objectives
* Subject has a history of non-response to an adequate (6-week) trial of 3 or more antidepressants (with or without mood stabilizers) during the current major depressive episode.
* Subject has any clinically significant unstable medical condition or any clinically significant chronic disease that would pose a risk to the subject or that might confound the results of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2021-12-21 (Actual); Primary Completion 2023-10-18 (Actual); Study Completion 2023-10-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CNS Medical Director, Study Chair — Sumitomo Pharma America, Inc.
Locations (89):
- United States (34):
  - University of Alabama at Birmingham Huntsville Regional Medical Campus, Huntsville, Alabama
  - Sanro Clinical Research Group LLC, Bryant, Arkansas
  - Advanced Research Center, Inc., Anaheim, California
  - Sun Valley Research Center, Imperial, California
  - Clinical innovations, Inc., Riverside, California
  - Siyan Clinical Research, Santa Rosa, California
  - Collaborative Neuroscience Research, LLC, Torrance, California
  - Vertex Research Group, Clermont, Florida
  - Sarkis Clinical Trials, Gainesville, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Premier Clinical Research Institute, Inc., Miami, Florida
  - Central Miami Medical Institute, Miami, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - GCP Clinical Research LLC, Tampa, Florida
  - Atlanta Behavioral Research, LLC, Atlanta, Georgia
  - Psych Atlanta, P.C., Marietta, Georgia
  - AMR Conventions Research, Warrenville, Illinois
  - Dept. of Psychiatry & Behavioral Sciences, University of Louisville School of Medicine, Louisville, Kentucky
  - St. Charles Psychiatric Associates / Midwest Research Group, Saint Charles, Missouri
  - Alivation Research, LLC, Lincoln, Nebraska
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - Global Medical Institutes, LLC, Princeton, New Jersey
  - UB Department of Psychiatry, Buffalo, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Richmond Behavioral Associates ERG Clinical Research - New York PLLC, Staten Island, New York
  - New Hope Clinical Research, Charlotte, North Carolina
  - Quest Therapeutics of Avon Lake, Avon Lake, Ohio
  - Neuro-Behavioral Clinical Research, Inc, North Canton, Ohio
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - Lehigh Center for Clinical Research, LLC, Allentown, Pennsylvania
  - Community Clinical Research, Inc., Austin, Texas
  - UTHealth Science Center at Houston, Houston, Texas
  - Family Psychiatry of The Woodlands, The Woodlands, Texas
  - Integrated Clinical Research, St. George, Utah
- Bulgaria (10):
  - State Psychiatric Hospital - Kardzhali First Women Department Third Men Department, Kardzhali
  - Medical Center Mentalcare OOD, Plovdiv
  - Mental Health Center- Ruse EOOD,Men Department for treatment of persons with acute psychotic disorders; Women Department for treatment of persons with acute psychotic disorders; Department "Daily stationary", Rousse
  - Mental Health Center - Sofia EOOD, Sofia
  - Medical Center Sveti Naum EOOD, Sofia
  - DCC St. Vrach and St. St. Kuzma and Damian OOD, Sofia
  - Medical Center Hera EOOD, Sofia
  - Medical Center Intermedica OOD, Sofia
  - State Psychiatric Hospital - s. Tsarev brod First Department for Active Treatment - Men Second Department for Active Treatment - Men Women Department - Rehabilitation Sector Women Department - Acute Sector, Tsarev Brod
  - DCC Mladost-M Varna OOD 15, Republika Blvd., MC Mladost, 3rd floor, Varna
- AMNDX Inc., Markham, Ontario, Canada
- Japan (35):
  - Hiro Mental Clinic, Fukuoka, Fukuoka
  - Shinseikai Kaku Mental Clinic, Fukuoka, Fukuoka
  - Mental Clinic Sakurazaka, Fukuoka, Fukuoka
  - Hatakeyama Clinic, Kitakyushu, Fukuoka
  - Someikai Kanagami Clinic, Kitakyushu-shi, Fukuoka
  - Kokura Mental Clinic, Kitakyushu-shi, Fukuoka
  - Hirota Clinic, Kurume-shi, Fukuoka
  - Shiranui Hospital, Omuta-shi, Fukuoka
  - Jisenkai Nanko Psychiatric Institute, Shirakawa-shi, Fukushima
  - Teine Keijinkai Hospital, Sapporo, Hokkaido
  - Tatsuta Clinic, Kobe, Hyōgo
  - Cerisier Heart Clinic, Kagoshima, Kagoshima-ken
  - Musashikosugi J Kokorono Clinic, Kawasaki-shi, Kanagawa
  - Yutaka Clinic, Sagamihara-shi, Kanagawa
  - Azamino Mental Clinic, Yokohama, Kanagawa
  - Yamatenomori Kokorono Clinic, Yokohama, Kanagawa
  - Satokai Yuge Hospital, Kumamoto, Kumamoto
  - Akari Clinic, Naha, Okinawa
  - Shiroma Clinic, Urasoe-shi, Okinawa
  - Rainbow & Sea Hospital, Karatsu-shi, Saga-ken
  - Juntendo University Hospital, Bunkyō City, Tokyo-To
  - Senzoku Psychosomatic Clinic, Meguro-ku, Tokyo-To
  - Minami-Aoyama Antique Street Clinic, Minatoku, Tokyo-To
  - Heart Care Ginga Clinic, Nakano, Tokyo-To
  - Sangenjaya Nakamura Mental Clinic, Setagaya-ku, Tokyo-To
  - Sangenjaya Neurology- Psychosomatic Clinic, Setagaya-ku, Tokyo-To
  - Japanese Red Cross Medical Center, Shibuya-ku, Tokyo-To
  - Maynds Tower Mental Clinic, Shibuya-ku, Tokyo-To
  - Sangubashi Kokorono Clinic, Shibuya-ku, Tokyo-To
  - Etoh Mental Clinic, Shinagawa-ku, Tokyo-To
  - Tamaki Clinic, Shinjuku-ku, Tokyo-To
  - Himorogi Psychiatric Institute, Shinjuku-ku, Tokyo-To
  - Uguisudani Mental Clinic, Taito-ku, Tokyo-To
  - Ohwa Mental Clinic, Toshima-ku, Tokyo-To
  - Kitaikebukuro Kokoro No Clinic, Toshima-ku, Tokyo-To
- Romania (7):
  - Spitalul Clinic de Psihiatrie si Neurologie Brasov, Sectia Psihiatrie Clinică I, Brasov
  - Spitalul Clinic de Psihiatrie ''Prof. Dr. Alexandru Obregia'', Bucharest
  - Spitalul Clinic de Psihiatrie, Bucharest
  - Sectia Psihiatrie, Centrul de Evaluare si Tratament al Toxicodependentelor pentru Tineri "Sfantul Stelian", Sectia Psihiatrie, Bucharest
  - Institutul Privat De Cercetări Melchisedec, Pentru Boli Autoimune, Ereditare Şi Rare - I.P.C.M., Craiova
  - Institutul de Psihiatrie Socola Iasi, Sectia Psihiatrie I Femei, Iași
  - Institutul de Psihiatrie Socola Iasi, Sectia Psihiatrie III Acuti, Iași
- Slovakia (2):
  - PsychoLine s. r. o., Psychiatricka ambulancia, Rimavská Sobota
  - Crystal Comfort s.r.o., Psychiatricka ambulancia, Vranov nad Topľou

IPD SHARING:
Plan to Share IPD: Yes
IPD for this study may be made available upon request via the Vivli Center for Global Clinical Research Data Site
Supporting Information: Study Protocol, SAP, CSR
Time Frame: IPD will be made available upon request within 12 months of posting the study results on ct.gov.
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.

REFERENCES:
- [Derived] Hopkins SC, Tomioka S, Szabo ST, Koblan KS. A clinical trial inclusion criteria to enrich for patients presenting with canonical symptom structure in bipolar depression. Contemp Clin Trials. 2024 Oct;145:107644. doi: 10.1016/j.cct.2024.107644. Epub 2024 Aug 3. PMID 39098761

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants had to go through at least 3 days or 5 half-lives antipsychotic medication washout.In total 83 Participants are Randomized in the trial, however one of the participant is randomized in error and was discontinued from study before taking any IP, So this subject is not considered in analysis population. Hence we have difference of 1 subject in Enrollment Number.
Period: Overall Study
Arm/Group | Placebo | SEP-4199 CR 200 mg | SEP-4199 CR 400 mg
Started | 27 | 27 | 28
Completed | 24 | 22 | 25
Not Completed | 3 | 5 | 3
Not completed — Adverse Event | 1 | 2 | 2
Not completed — Lost to Follow-up | 0 | 0 | 1
Not completed — Withdrawal by Subject | 2 | 1 | 0
Not completed — Other Study Discontinuation Reason | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | SEP-4199 CR 200 mg | SEP-4199 CR 400 mg | Total
Number analyzed (Participants) | 27 | 27 | 28 | 82
Age, Continuous [Mean (Standard Deviation); unit: Years] | 43.9 (11.34) | 46.7 (11.67) | 42.8 (12.53) | 44.5 (11.83)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 17 | 17 | 52
  Male | 9 | 10 | 11 | 30
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 10 | 9 | 10 | 29
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 2 | 3
  White | 16 | 18 | 16 | 50
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6 | 5 | 7 | 18
  Bulgaria | 11 | 12 | 11 | 34
  Romania | 0 | 1 | 0 | 1
  Japan | 10 | 9 | 10 | 29
Baseline Montgomery-Asberg Depression Rating Scale( MADRS )Total Score [Mean (Standard Deviation); unit: units on a scale] — Montgomery-Asberg Depression Rating Scale( MADRS ) is a clinician-rated assessment of the subject's level of depression. The measure contains 10 items that measure apparent and reported sadness, inner tension, reduced sleep and appetite, difficulty concentrating, lassitude, inability to feel, and pessimistic and suicidal thoughts, each ranging from 0 to 6. The MADRS total score ranges from 0 to 60, with higher scores indicating increased depressive symptoms
  units on a scale | 36.6 (5.64) | 37.5 (6.22) | 37.6 (4.92) | 37.2 (5.55)
Baseline Clinical Global Impressions - Severity: Bipolar Version (CGI-BP-S) score (depression) [Mean (Standard Deviation); unit: units on a scale] — Clinical Global Impressions - Severity: Bipolar Version (CGI-BP-S) score (depression) is a single value, clinician-rated assessment of illness severity, and 7-point scale with range from 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; 7 = among the most extremely ill subjects. A higher score is associated with greater illness severity.
  units on a scale | 5 (0.65) | 5 (0.68) | 4.9 (0.69) | 5 (0.66)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Montgomery-Asberg Depression Rating Scale (MADRS) Total Score at Week 6
Description: Montgomery-Asberg Depression Rating Scale (MADRS) is a clinician-rated assessment of the subject's level of depression. The measure contains 10 items that measure apparent and reported sadness, inner tension, reduced sleep and appetite, difficulty concentrating, lassitude, inability to feel, and pessimistic and suicidal thoughts, each ranging from 0 to 6. The MADRS total score ranges from 0 to 60, with higher scores indicating increased depressive symptoms
Time Frame: 6 Weeks
Population: ITT population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | SEP-4199 CR 200 mg | SEP-4199 CR 400 mg
Number analyzed (Participants) | 27 | 27 | 28
units on a scale | -10.33 (2.004) | -14.27 (2.055) | -16.67 (2.014)
Statistical Analysis 1: Comparison: Placebo vs SEP-4199 CR 200 mg; Test type: Superiority; p = 0.1718, Mixed Models Analysis; Mean Difference (Final Values) = -3.94, 95% CI 2-sided [-9.64 to 1.75], Standard Error of Mean 2.857
Statistical Analysis 2: Comparison: Placebo vs SEP-4199 CR 400 mg; Test type: Superiority; p = 0.028600, Mixed Models Analysis; Mean Difference (Final Values) = -6.34, 95% CI 2-sided [-11.99 to -0.68], Standard Error of Mean 2.837

2. Secondary Outcome: Change From Baseline in Global Severity Assessed by the Clinical Global Impressions Severity: Bipolar Version (CGI-BP-S) Score (Depression) at Week 6
Description: Clinical Global Impressions Severity: Bipolar Version (CGI-BP-S) score (depression) is a single value, clinician-rated assessment of illness severity, and 7-point scale with range from 1 = normal, not at all ill; 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; 7 = among the most extremely ill subjects. A higher score is associated with greater illness severity.
Time Frame: 6 Weeks
Population: ITT population
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | SEP-4199 CR 200 mg | SEP-4199 CR 400 mg
Number analyzed (Participants) | 27 | 27 | 28
units on a scale | -1.16 (0.214) | -1.26 (0.222) | -1.46 (0.217)
Statistical Analysis 1: Comparison: Placebo vs SEP-4199 CR 200 mg; Test type: Superiority; p = 0.7314, Mixed Models Analysis; Mean Difference (Final Values) = -0.11, 95% CI 2-sided [-0.72 to 0.51], Standard Error of Mean 0.308
Statistical Analysis 2: Comparison: Placebo vs SEP-4199 CR 400 mg; Test type: Superiority; p = 0.3169, Mixed Models Analysis; Mean Difference (Final Values) = -0.31, 95% CI 2-sided [-0.91 to 0.3], Standard Error of Mean 0.305

ADVERSE EVENTS:
Time Frame: Up to 7 weeks
Description: Adverse events were untoward medical occurrences that occurred on or after the first dose of study medication.
Arm/Group | Placebo | SEP-4199 CR 200 mg | SEP-4199 CR 400 mg
All-Cause Mortality (participants affected / at risk) | 0/27 | 0/27 | 0/28
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/27 | 0/28
Other Adverse Events (participants affected / at risk) | 7/27 | 1/27 | 6/28
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=27) | SEP-4199 CR 200 mg (N=27) | SEP-4199 CR 400 mg (N=28)
Somnolence (Nervous system disorders) | 2 (2) | 0 (0) | 2 (3)
Headache (Nervous system disorders) | 3 (4) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0) | 2 (2)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish.

DOCUMENTS (2):
  • Study Protocol (2022-12-06): https://cdn.clinicaltrials.gov/large-docs/10/NCT05169710/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-08): https://cdn.clinicaltrials.gov/large-docs/10/NCT05169710/SAP_001.pdf